CLINICAL TRIAL: NCT03170609
Title: A PHASE 1/2, RANDOMIZED, PLACEBO-CONTROLLED, OBSERVER-BLINDED TRIAL TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A MULTIVALENT GROUP B STREPTOCOCCUS VACCINE IN HEALTHY ADULTS 18 TO 49 YEARS OF AGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: C1091001
Record Dates: First submitted 2017-05-26; First posted 2017-05-31 (Actual); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Group B Streptococcal Infections
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (7):
- Lowest dose formulation a (Experimental): Multivalent group B streptococcus vaccine
  Interventions: Biological: Multivalent group B streptococcus vaccine
- Middle dose formulation a (Experimental): Multivalent group B streptococcus vaccine
  Interventions: Biological: Multivalent group B streptococcus vaccine
- Highest dose formulation a (Experimental): Multivalent group B streptococcus vaccine
  Interventions: Biological: Multivalent group B streptococcus vaccine
- Lowest dose formulation b (Experimental): Multivalent group B streptococcus vaccine
  Interventions: Biological: Multivalent group B streptococcus vaccine
- Middle dose formulation b (Experimental): Multivalent group B streptococcus vaccine
  Interventions: Biological: Multivalent group B streptococcus vaccine
- Highest dose formulation b (Experimental): Multivalent group B streptococcus vaccine
  Interventions: Biological: Multivalent group B streptococcus vaccine
- Placebo (Placebo Comparator): Saline control
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Multivalent group B streptococcus vaccine — Various formulations at three dose levels
  Arms: Highest dose formulation a; Highest dose formulation b; Lowest dose formulation a; Lowest dose formulation b; Middle dose formulation a; Middle dose formulation b
Biological: Placebo — Saline Control
  Arms: Placebo

SUMMARY:
This is the Phase 1/2 first-in-human, randomized, placebo-controlled, observer-blinded study evaluating the investigational multivalent group B streptococcus vaccine. Healthy adults aged 18 to 49 years of age with no history of group B streptococcal vaccination will be randomized to receive either a single intramuscular dose of multivalent group B streptococcus vaccine (various formulations at 3 dose levels) or a placebo (saline control).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults (male and female) 18 to 49 years of age at enrollment who are determined by medical history, physical examination, and clinical judgment of the investigator to be eligible for inclusion in the study.
2. Negative urine pregnancy test at Visit 1 for all female subjects who are of childbearing potential.

Exclusion Criteria:

1. Male subjects and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for at least 3 months after the last dose of investigational product.
2. Acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study. Chronic medical conditions include human immunodeficiency virus, chronic hepatitis B virus (HBV) infection (HBV surface antigen positive), and/or hepatitis C virus infection.
3. History of severe adverse reaction and/or severe allergic reaction (eg, anaphylaxis) to any vaccine.
4. History of microbiologically proven invasive disease caused by group B streptococcus (Streptococcus agalactiae).
5. Previous vaccination with any licensed or investigational group B streptococcus vaccine, or planned receipt during the subject's participation in the study (through the last blood draw).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2017-06-05 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Kentucky Pediatric / Adult Research, Bardstown, Kentucky
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Absalon J, Segall N, Block SL, Center KJ, Scully IL, Giardina PC, Peterson J, Watson WJ, Gruber WC, Jansen KU, Peng Y, Munson S, Pavliakova D, Scott DA, Anderson AS. Safety and immunogenicity of a novel hexavalent group B streptococcus conjugate vaccine in healthy, non-pregnant adults: a phase 1/2, randomised, placebo-controlled, observer-blinded, dose-escalation trial. Lancet Infect Dis. 2021 Feb;21(2):263-274. doi: 10.1016/S1473-3099(20)30478-3. Epub 2020 Sep 3. PMID 32891191
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1091001&StudyName=A+Phase+1%2C+Randomized%2C+Observer+Blinded+Trial+To+Evaluate+The+Safety%2C+Tolerability%2C+And+Immunogenicity+Of+A+Multivalent+Group+B+Streptococcus+Vaccine+In+Healthy+Adults+Aged+18+To+49+Years
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1091001&StudyName=A+Phase+1%2F2%2C+Randomized%2C+Placebo-controlled%2C+Observer-blinded+Trial+To+Evaluate+The+Safety%2C+Tolerability%2C+And+Immunogenicity+Of+A+Multivalent+Group+B+Streptococcus+Vaccine+In+Healthy+Adults+18+To+49+Years+Of+Age

RESULTS

PARTICIPANT FLOW:
Groups:
- GBS6 5 Microgram With Aluminum Phosphate: Participants were randomized to receive a single dose of 5 microgram of Group B Streptococcus 6-valent (GBS6) vaccine with aluminium phosphate, intramuscularly on Day 1 and were followed up to 6 months.
- GBS6 5 Microgram Without Aluminum Phosphate: Participants were randomized to receive a single dose of 5 microgram of GBS6 vaccine without aluminium phosphate, intramuscularly on Day 1 and were followed up to 6 months.
- GBS6 10 Microgram With Aluminum Phosphate: Participants were randomized to receive a single dose of 10 microgram of GBS6 vaccine with aluminium phosphate, intramuscularly on Day 1 and were followed up to 6 months.
- GBS6 10 Microgram Without Aluminum Phosphate: Participants were randomized to receive a single dose of 10 microgram of GBS6 vaccine without aluminium phosphate, intramuscularly on Day 1 and were followed up to 6 months.
- GBS6 20 Microgram With Aluminum Phosphate: Participants were randomized to receive a single dose of 20 microgram of GBS6 vaccine with aluminium phosphate, intramuscularly on Day 1 and were followed up to 6 months.
- GBS6 20 Microgram Without Aluminum Phosphate: Participants were randomized to receive a single dose of 20 microgram of GBS6 vaccine without aluminium phosphate, intramuscularly on Day 1 and were followed up to 6 months.
- Placebo: Participants were randomized to receive placebo (saline control) intramuscularly on Day 1 and were followed up to 6 months.
Period: Overall Study
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
Started | 53 | 52 | 52 | 52 | 52 | 52 | 52
Vaccinated | 52 | 52 | 52 | 52 | 52 | 52 | 52
Completed | 50 | 50 | 46 | 50 | 51 | 50 | 51
Not Completed | 3 | 2 | 6 | 2 | 1 | 2 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 5 | 2 | 1 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received either GBS6 vaccine or placebo.
Groups:
- GBS6 5 Microgram With Aluminum Phosphate: Participants were randomized to receive a single dose of 5 microgram of GBS6 vaccine with aluminium phosphate, intramuscularly on Day 1 and were followed up to 6 months.
- Total: Total of all reporting groups
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo | Total
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52 | 52 | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (8.43) | 34.7 (9.35) | 32.8 (8.31) | 31.9 (8.10) | 33.2 (8.67) | 30.5 (8.25) | 32.8 (8.74) | 32.7 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 41 | 32 | 33 | 35 | 37 | 43 | 256
  Male | 17 | 11 | 20 | 19 | 17 | 15 | 9 | 108
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 2 | 2 | 5 | 1 | 5 | 21
  Not Hispanic or Latino | 50 | 47 | 50 | 49 | 47 | 51 | 47 | 341
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 41 | 46 | 41 | 45 | 46 | 44 | 307
  Black or African American | 5 | 9 | 5 | 8 | 4 | 4 | 7 | 42
  Other | 2 | 1 | 0 | 2 | 2 | 2 | 0 | 9
  Asian | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 5
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Laboratory Abnormalities at 1-Week After Vaccination as Measured by Food and Drug Administration (FDA) Grade
Description: Hemoglobin:Grade(G)1: 11-13.5g/dL, G2:9.5-12.4g/dL,G3:8-10.4 g/dL, G4:<8.0 g/dL; leukocyte increase:G1: 10.8-15*10^9/Liter[L],G2:>15-20*10^9/L, G3:>20-25*10^9/L, G4:>25*10^9/L,leukocyte decrease: G1: 2.5-3.5*10^9/L, G2: 1.5-<2.5*10^9/L, G3: 1-<1.5*10^9/L, G4:<1*10^9/L; neutrophil decrease:G1: 1.5-2*10^9/L, G2:1-<1.5*10^9/L, G3:0.5-<1*10^9/L,G4:<0.5*10^9/L; platelets:G1: 125-140*10^9/L, G2:100-124*10^9/L, G3:25-99*10^9/L, G4:<25*10^9/L; eosinophils: G1: 0.65-1.5*10^9/L, G2:>1.5-5*10^9/L, G3:>5*10^9/L, G4: hypereosinophilic;alanine aminotransferase,aspartate aminotransferase:G1: 1.1-2.5 *ULN, G2:2.6-5.0*ULN, G3:5.1-10*ULN, G4:>10*ULN; alkaline phosphatase:G1: 1.1-2*ULN, G2:2.1-3*ULN, G3:3.1-10*ULN, G4:>10*ULN; Bilirubin:G1: 1.1-1.5*ULN, G2: 1.26-2*ULN,G3: 1.51-3.0*ULN,G4:>1.75*ULN;blood urea nitrogen:G1:23-26mg/dL,G2:27-31mg/dL,G3:>31mg/dL, G4:dialysis;creatinine:G1:1.5-1.7mg/dL,G2:1.8-2mg/dL,G3:2.1-2.5 mg/dL,G4:dialysis.Categories with>=1 participant with abnormality are reported only.
Time Frame: 1 week after vaccination
Population: Analysis population for this outcome measure included a subset of participants who received GBS6 vaccine or placebo.
Measure: Number; unit: percentage of participants
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16 | 24
percentage of participants
  Hemoglobin: Grade 1 | 0 | 6.3 | 12.5 | 0 | 0 | 6.3 | 0
  Hemoglobin: Grade 2 | 6.3 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets: Grade 1 | 0 | 0 | 6.3 | 6.7 | 0 | 0 | 0
  Leukocyte decrease:Grade 1 | 6.3 | 6.3 | 0 | 0 | 0 | 0 | 0
  Leukocyte increase: Grade 1 | 0 | 0 | 0 | 0 | 0 | 6.3 | 0
  Leukocyte increase: Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 4.2
  Neutrophils decrease(Absolute): Grade 1 | 6.3 | 18.8 | 0 | 0 | 0 | 6.3 | 0
  Neutrophils decrease (Absolute): Grade 2 | 0 | 0 | 0 | 0 | 6.3 | 0 | 0
  Blood urea nitrogen: Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4.2
  Blood urea nitrogen: Grade 2 | 0 | 0 | 0 | 0 | 0 | 6.3 | 0
  Aspartate aminotransferase: Grade 1 | 0 | 0 | 0 | 0 | 6.3 | 0 | 0
  Aspartate aminotransferase: Grade 3 | 0 | 6.3 | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase: Grade 1 | 0 | 6.3 | 0 | 0 | 12.5 | 0 | 0
  Bilirubin in presence of normal AST and ALT:Grade1 | 0 | 0 | 6.3 | 0 | 0 | 0 | 0
  Alkaline phosphate: Grade 1 | 0 | 0 | 6.3 | 0 | 0 | 0 | 0

2. Primary Outcome: Percentage of Participants With Local Reactions by Maximum Severity Within 14 Days After Vaccination
Description: Local reactions were collected by using an e-diary and included redness, swelling and pain at injection site. Redness and swelling were graded as: mild (2.5-5.0 centimeter [cm]), moderate (greater than [>] 5.0-10.0 cm) and severe (>10.0 cm), grade 4 for redness (necrosis or exfoliative dermatitis) and grade 4 for swelling (necrosis). Pain at injection site was graded as: mild (did not interfere with activity), moderate (repeated use of nonnarcotic pain reliever >24 hours or interfered with activity), severe (any use of narcotic pain reliever or prevented daily activity which resulted in missed days of work or school or was otherwise incapacitating, or included use of narcotics for analgesia), and grade 4 (required emergency room visit or hospitalization). The maximum severity (highest grading) of each location reaction within 14 days of vaccination was derived.
Time Frame: Within 14 days after vaccination
Population: Safety population included all participants who received GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52 | 52
percentage of participants
  Pain:Any | 53.8 [39.5 to 67.8] | 32.7 [20.3 to 47.1] | 48.1 [34.0 to 62.4] | 38.5 [25.3 to 53.0] | 51.9 [37.6 to 66.0] | 25.0 [14.0 to 38.9] | 15.4 [6.9 to 28.1]
  Pain:Mild | 51.9 [37.6 to 66.0] | 28.8 [17.1 to 43.1] | 44.2 [30.5 to 58.7] | 36.5 [23.6 to 51.0] | 42.3 [28.7 to 56.8] | 19.2 [9.6 to 32.5] | 13.5 [5.6 to 25.8]
  Pain:Moderate | 1.9 [0.0 to 10.3] | 3.8 [0.5 to 13.2] | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.3] | 9.6 [3.2 to 21.0] | 5.8 [1.2 to 15.9] | 1.9 [0.0 to 10.3]
  Pain:Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Pain:Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Redness:Any | 0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 5.8 [1.2 to 15.9] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Redness:Mild | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 5.8 [1.2 to 15.9] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Redness:Moderate | 0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Redness:Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Redness:Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Swelling:Any | 0 [0.0 to 6.8] | 5.8 [1.2 to 15.9] | 1.9 [0.0 to 10.3] | 3.8 [0.5 to 13.2] | 5.8 [1.2 to 15.9] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Swelling:Mild | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.3] | 3.8 [0.5 to 13.2] | 5.8 [1.2 to 15.9] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Swelling:Moderate | 0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Swelling:Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Swelling:Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]

3. Primary Outcome: Percentage of Participants With Systemic Events by Maximum Severity Within 14 Days After Vaccination
Description: Fever:38.0-38.4 degree Celsius (C),38.5-38.9 degree C,39.0-40.0 degree C,>40.0 degree C;nausea/vomiting:mild(not interfered with activity/1-2times in 24 hours[hr]),moderate(some interference with activity/>2times in 24hr),severe(prevented daily activity;required intravenous hydration); diarrhea:mild(2-3 loose stools in 24hr),moderate(4-5 loose stools in 24hr),severe(>=6 loose stools in 24 hr); headache:mild(not interfered with activity),moderate(repeated use of non-narcotic pain reliever >24 hr/some interference with activity),severe(significant;any use of narcotic pain reliever/prevented daily activity);fatigue,muscle and joint pain:mild(not interfered with activity), moderate(some interference with activity),severe(significant;prevented daily activity).Prevented daily activity=missed days of work, school/otherwise incapacitating/use of narcotics for analgesia.Nausea/vomiting,diarrhea,headache,fatigue/tiredness,muscle and joint pain: grade 4=emergency room visit or hospitalization.
Time Frame: Within 14 days after vaccination
Population: Safety population included all participants who received GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52 | 52
percentage of participants
  Fever:>=38.0 degree C | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.3]
  Fever:38.0 to 38.4 degree C | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8]
  Fever:38.5 to 38.9 degree C | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3]
  Fever:39.0 to 40.0 degree C | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Fever:>40.0 degree C | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Nausea/vomiting: Any | 13.5 [5.6 to 25.8] | 5.8 [1.2 to 15.9] | 11.5 [4.4 to 23.4] | 17.3 [8.2 to 30.3] | 9.6 [3.2 to 21.0] | 11.5 [4.4 to 23.4] | 21.2 [11.1 to 34.7]
  Nausea/vomiting: Mild | 9.6 [3.2 to 21.0] | 3.8 [0.5 to 13.2] | 9.6 [3.2 to 21.0] | 11.5 [4.4 to 23.4] | 7.7 [2.1 to 18.5] | 9.6 [3.2 to 21.0] | 13.5 [5.6 to 25.8]
  Nausea/vomiting: Moderate | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.3] | 5.8 [1.2 to 15.9] | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.3] | 7.7 [2.1 to 18.5]
  Nausea/vomiting: Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Nausea/vomiting: Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Diarrhea:Any | 13.5 [5.6 to 25.8] | 21.2 [11.1 to 34.7] | 13.5 [5.6 to 25.8] | 21.2 [11.1 to 34.7] | 21.2 [11.1 to 34.7] | 17.3 [8.2 to 30.3] | 11.5 [4.4 to 23.4]
  Diarrhea:Mild | 11.5 [4.4 to 23.4] | 21.2 [11.1 to 34.7] | 11.5 [4.4 to 23.4] | 13.5 [5.6 to 25.8] | 19.2 [9.6 to 32.5] | 11.5 [4.4 to 23.4] | 5.8 [1.2 to 15.9]
  Diarrhea:Moderate | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 3.8 [0.5 to 13.2] | 0 [0.0 to 6.8] | 5.8 [1.2 to 15.9] | 5.8 [1.2 to 15.9]
  Diarrhea:Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Diarrhea:Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Headache:Any | 40.4 [27.0 to 54.9] | 36.5 [23.6 to 51.0] | 32.7 [20.3 to 47.1] | 38.5 [25.3 to 53.0] | 40.4 [27.0 to 54.9] | 30.8 [18.7 to 45.1] | 42.3 [28.7 to 56.8]
  Headache:Mild | 26.9 [15.6 to 41.0] | 21.2 [11.1 to 34.7] | 15.4 [6.9 to 28.1] | 11.5 [4.4 to 23.4] | 28.8 [17.1 to 43.1] | 11.5 [4.4 to 23.4] | 23.1 [12.5 to 36.8]
  Headache:Moderate | 13.5 [5.6 to 25.8] | 13.5 [5.6 to 25.8] | 15.4 [6.9 to 28.1] | 25.0 [14.0 to 38.9] | 11.5 [4.4 to 23.4] | 17.3 [8.2 to 30.3] | 15.4 [6.9 to 28.1]
  Headache:Severe | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.3] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 3.8 [0.5 to 13.2]
  Headache:Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Fatigue/tiredness: Any | 42.3 [28.7 to 56.8] | 32.7 [20.3 to 47.1] | 34.6 [22.0 to 49.1] | 26.9 [15.6 to 41.0] | 50.0 [35.8 to 64.2] | 38.5 [25.3 to 53.0] | 34.6 [22.0 to 49.1]
  Fatigue/tiredness: Mild | 19.2 [9.6 to 32.5] | 11.5 [4.4 to 23.4] | 9.6 [3.2 to 21.0] | 7.7 [2.1 to 18.5] | 25.0 [14.0 to 38.9] | 19.2 [9.6 to 32.5] | 9.6 [3.2 to 21.0]
  Fatigue/tiredness: Moderate | 23.1 [12.5 to 36.8] | 21.2 [11.1 to 34.7] | 21.2 [11.1 to 34.7] | 15.4 [6.9 to 28.1] | 25.0 [14.0 to 38.9] | 19.2 [9.6 to 32.5] | 19.2 [9.6 to 32.5]
  Fatigue/tiredness: Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 3.8 [0.5 to 13.2] | 3.8 [0.5 to 13.2] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 5.8 [1.2 to 15.9]
  Fatigue/tiredness:Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Muscle pain:Any | 17.3 [8.2 to 30.3] | 25.0 [14.0 to 38.9] | 19.2 [9.6 to 32.5] | 19.2 [9.6 to 32.5] | 19.2 [9.6 to 32.5] | 23.1 [12.5 to 36.8] | 19.2 [9.6 to 32.5]
  Muscle pain:Mild | 9.6 [3.2 to 21.0] | 17.3 [8.2 to 30.3] | 7.7 [2.1 to 18.5] | 11.5 [4.4 to 23.4] | 13.5 [5.6 to 25.8] | 17.3 [8.2 to 30.3] | 5.8 [1.2 to 15.9]
  Muscle pain:Moderate | 7.7 [2.1 to 18.5] | 7.7 [2.1 to 18.5] | 9.6 [3.2 to 21.0] | 7.7 [2.1 to 18.5] | 5.8 [1.2 to 15.9] | 5.8 [1.2 to 15.9] | 11.5 [4.4 to 23.4]
  Muscle pain:Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0.0 [0.0 to 6.8] | 1.9 [0.0 to 10.3]
  Muscle pain:Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Joint pain:Any | 13.5 [5.6 to 25.8] | 9.6 [3.2 to 21.0] | 13.5 [5.6 to 25.8] | 9.6 [3.2 to 21.0] | 13.5 [5.6 to 25.8] | 11.5 [4.4 to 23.4] | 5.8 [1.2 to 15.9]
  Joint pain:Mild | 9.6 [3.2 to 21.0] | 5.8 [1.2 to 15.9] | 3.8 [0.5 to 13.2] | 7.7 [2.1 to 18.5] | 9.6 [3.2 to 21.0] | 9.6 [3.2 to 21.0] | 1.9 [0.0 to 10.3]
  Joint pain:Moderate | 3.8 [0.5 to 13.2] | 3.8 [0.5 to 13.2] | 9.6 [3.2 to 21.0] | 1.9 [0.0 to 10.3] | 3.8 [0.5 to 13.2] | 1.9 [0.0 to 10.3] | 3.8 [0.5 to 13.2]
  Joint pain:Severe | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]
  Joint pain:Grade 4 | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]

4. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or that was considered to be an important medical event. AEs included both non-serious AEs and SAEs.
Time Frame: Within 1 month after vaccination
Population: Safety population included all participants who received GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52 | 52
percentage of participants | 19.2 [9.6 to 32.5] | 5.8 [1.2 to 15.9] | 19.2 [9.6 to 32.5] | 13.5 [5.6 to 25.8] | 26.9 [15.6 to 41.0] | 28.8 [17.1 to 43.1] | 21.2 [11.1 to 34.7]

5. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) Within 6 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or that was considered to be an important medical event.
Time Frame: Within 6 months after vaccination
Population: Safety population included all participants who received GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52 | 52
percentage of participants | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 1.9 [0.0 to 10.3] | 0 [0.0 to 6.8] | 0 [0.0 to 6.8]

6. Primary Outcome: Percentage of Participants With Medically Attended Adverse Events (MAEs) Within 6 Months After Vaccination
Description: An AE was any untoward medical occurrence in a participant in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly or that was considered to be an important medical event. An MAE was defined as a non serious AE (AE other than SAE) that resulted in an evaluation at a medical facility.
Time Frame: Within 6 months after vaccination
Population: Safety population included all participants who received GBS6 vaccine or placebo.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
Number analyzed (Participants) | 52 | 52 | 52 | 52 | 52 | 52 | 52
percentage of participants | 21.2 [11.1 to 34.7] | 23.1 [12.5 to 36.8] | 28.8 [17.1 to 43.1] | 19.2 [9.6 to 32.5] | 34.6 [22.0 to 49.1] | 26.9 [15.6 to 41.0] | 34.6 [22.0 to 49.1]

7. Secondary Outcome: GBS6 Serotype-Specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) at 1 Month After Vaccination
Description: Serotypes used for evaluation were: Ia, Ib, II, III, IV, and V.
Time Frame: 1 month after vaccination
Population: Evaluable immunogenicity population included all eligible participants who received GBS6 vaccine or placebo, had 1 month after vaccination blood drawn for assay and had at least 1 valid determinate assay result with no major protocol violation. 'Number analyzed' = number of participants with valid, determinate assay results for specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: Microgram per milliliter
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
Number analyzed (Participants) | 51 | 51 | 51 | 50 | 52 | 52 | 47
Microgram per milliliter
  Ia: number analyzed (Participants) | 51 | 50 | 51 | 50 | 52 | 52 | 47
  Ia | 30.880 [13.301 to 71.691] | 20.341 [8.533 to 48.486] | 24.723 [10.577 to 57.785] | 41.826 [17.740 to 98.613] | 21.125 [10.121 to 44.094] | 17.829 [7.542 to 42.149] | 0.755 [0.372 to 1.536]
  Ib: number analyzed (Participants) | 51 | 51 | 51 | 49 | 52 | 52 | 47
  Ib | 2.060 [0.891 to 4.762] | 2.051 [0.952 to 4.417] | 3.174 [1.368 to 7.365] | 3.639 [1.426 to 9.289] | 2.742 [1.102 to 6.820] | 1.948 [0.785 to 4.836] | 0.034 [0.019 to 0.059]
  II | 31.851 [17.303 to 58.630] | 21.919 [11.544 to 41.618] | 26.980 [14.586 to 49.904] | 57.011 [31.917 to 101.832] | 37.258 [20.764 to 66.853] | 31.786 [17.490 to 57.770] | 0.187 [0.126 to 0.279]
  III: number analyzed (Participants) | 51 | 51 | 50 | 49 | 52 | 52 | 47
  III | 5.683 [3.002 to 10.760] | 4.531 [2.290 to 8.965] | 4.979 [2.346 to 10.571] | 12.806 [6.221 to 26.365] | 5.559 [2.724 to 11.345] | 3.766 [1.887 to 7.517] | 0.081 [0.054 to 0.122]
  IV | 2.915 [1.712 to 4.964] | 5.149 [2.913 to 9.102] | 4.924 [3.077 to 7.879] | 4.908 [2.890 to 8.336] | 4.303 [2.605 to 7.107] | 7.018 [4.518 to 10.903] | 0.046 [0.027 to 0.078]
  V | 2.985 [1.346 to 6.619] | 3.368 [1.477 to 7.679] | 4.702 [2.033 to 10.878] | 5.142 [2.403 to 11.005] | 3.991 [1.984 to 8.031] | 6.760 [3.230 to 14.146] | 0.143 [0.084 to 0.244]

ADVERSE EVENTS:
Time Frame: Local reactions and systemic events: within 14 days after vaccination on Day 1 and all AEs other than local reactions and systemic events: within 6 Months after vaccination on Day 1
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.Safety population included all participants who received GBS6 vaccine or placebo.
Arm/Group | GBS6 5 Microgram With Aluminum Phosphate | GBS6 5 Microgram Without Aluminum Phosphate | GBS6 10 Microgram With Aluminum Phosphate | GBS6 10 Microgram Without Aluminum Phosphate | GBS6 20 Microgram With Aluminum Phosphate | GBS6 20 Microgram Without Aluminum Phosphate | Placebo
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 1/52 | 0/52 | 0/52 | 0/52 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52 | 0/52 | 1/52 | 0/52 | 1/52 | 0/52 | 0/52
Other Adverse Events (participants affected / at risk) | 40/52 | 35/52 | 39/52 | 36/52 | 41/52 | 36/52 | 35/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBS6 5 Microgram With Aluminum Phosphate (N=52) | GBS6 5 Microgram Without Aluminum Phosphate (N=52) | GBS6 10 Microgram With Aluminum Phosphate (N=52) | GBS6 10 Microgram Without Aluminum Phosphate (N=52) | GBS6 20 Microgram With Aluminum Phosphate (N=52) | GBS6 20 Microgram Without Aluminum Phosphate (N=52) | Placebo (N=52)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GBS6 5 Microgram With Aluminum Phosphate (N=52) | GBS6 5 Microgram Without Aluminum Phosphate (N=52) | GBS6 10 Microgram With Aluminum Phosphate (N=52) | GBS6 10 Microgram Without Aluminum Phosphate (N=52) | GBS6 20 Microgram With Aluminum Phosphate (N=52) | GBS6 20 Microgram Without Aluminum Phosphate (N=52) | Placebo (N=52)
Diarrhoea (Gastrointestinal disorders) | 7 | 11 | 7 | 11 | 11 | 9 | 6
Nausea/vomiting (Gastrointestinal disorders) | 7 | 3 | 6 | 9 | 5 | 6 | 11
Fatigue (General disorders) | 22 | 17 | 18 | 14 | 26 | 20 | 18
Influenza (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 0 | 1 | 3 | 2
Sinusitis (Infections and infestations) | 4 | 2 | 2 | 1 | 2 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 3 | 1 | 4 | 6 | 3
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 7 | 5 | 7 | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 13 | 10 | 10 | 10 | 12 | 10
Headache (Nervous system disorders) | 21 | 19 | 17 | 20 | 21 | 16 | 22
Migraine (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 3
Injection site pain (General disorders) | 28 | 17 | 25 | 20 | 27 | 13 | 8
Injection site swelling (General disorders) | 0 | 3 | 1 | 2 | 3 | 0 | 0
Injection site erythema (General disorders) | 0 | 2 | 1 | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT03170609/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT03170609/SAP_001.pdf